CLINICAL TRIAL: NCT02041182
Title: Use of an Electronic Pre-visit Questionnaire and Effect on Patient-provider Discussions of Youth Violence in Primary Care
Brief Title: Electronic Pre-visit Questionnaire to Prompt Discussions of Youth Violence in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: APA-YIA-2013
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-01

CONDITIONS: Exposure to Violent Event; Bullying
Keywords: youth violence; doctor-patient communication; health risk behaviors; pre-visit questionnaires
MeSH Terms: conditions — Bullying; Health Risk Behaviors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Pre-visit Questionnaire (Experimental): Adolescents receive PVQ that includes questions about youth violence/bullying
  Interventions: Behavioral: Pre-Visit Questionnaire
- Control Pre-visit Questionnaire (Active Comparator): Adolescents received PVQ without youth violence/bullying items
  Interventions: Behavioral: Pre-Visit Questionnaire

INTERVENTIONS:
Behavioral: Pre-Visit Questionnaire

SUMMARY:
Pediatricians are supposed to talk about youth violence at all heath supervision visits, however these types of conversations rarely occur. There have been no studies assessing tools to prompt these discussions. The goal of this study is to see if electronic pre-visit questionnaires (PVQs) prompt patient-provider discussion of youth violence (YV) in the primary care setting. Additionally, patient-provider characteristics are explored as mediators to youth violence discussions, as well as feasibility and acceptability of the PVQ by patients and providers.

Adolescents ages 13 to 21 who come to the Hasbro Primary Care Clinics for annual physicals will be recruited. A baseline phase was conducted to look at how often providers ask about health-related teen behaviors, assessed by exit survey. The experimental period will involve adolescents completing health-related behavior PVQ, given to their doctor prior to the visit. Exit survey will assess topics discussed. Experimental group will differ from control group based on PVQ containing extra questions about youth violence.

ELIGIBILITY:
Inclusion Criteria:

* adolescents ages 13-21
* presenting for annual physical exam
* provider is general pediatrician (micro-practice 1-8)
* parent present for consent (if under 18 years old)

Exclusion Criteria:

* non-English speaking
* developmental/neurologic delay
* no parent (if under 18 years old)
* presenting for sick visit or specialty clinic

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of patient-reported patient-provider discussions about youth violence | One time point (single day)
  The intervention is implemented immediately prior to the primary care visit; the outcome is measured directly following the visit by exit survey

CONTACTS AND LOCATIONS:
Overall Officials: Megan Ranney, MD MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Primary Care Clinics, Providence, Rhode Island, United States